CLINICAL TRIAL: NCT01585129
Title: Treatment Utility of Postpartum Antibiotics in Chorioamnionitis
Acronym: TUPAC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility in patient enrollment
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0704
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: The Primary Outcome of This Study Will be the Rate of Endometritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postpartum Antibiotics (Experimental): Patients will receive one additional dose of postpartum antibiotics (Clinda, Gentamicin)
  Interventions: Drug: Postpartum Antibiotics
- No postpartum antibiotics (Placebo Comparator): No further postpartum antibiotics
  Interventions: Drug: No postpartum antibiotics

INTERVENTIONS:
Drug: Postpartum Antibiotics — Patients randomized into this arm will receive one additional dose of gentamicin (1.5 mg/kg) and clindamycin (900mg) in the postpartum setting.
  Arms: Postpartum Antibiotics
Drug: No postpartum antibiotics — Patients randomized into this arm will not receive any postpartum antibiotics after delivery. They will be managed identically to the other arm in terms of chorioamnionitis (fever pre-delivery). The groups will be managed identically if endometritis (post-partum fever) develops.
  Arms: No postpartum antibiotics

SUMMARY:
To determine if prophylactic postpartum antibiotics are required post-cesarean delivery for pregnancies with treated chorioamnionitis.

DETAILED DESCRIPTION:
Bacterial infection of the amniotic cavity, termed "chorioamnionitis", is a major cause of perinatal mortality and maternal morbidity. Early administration of broad-spectrum antibiotic therapy in the laboring patient with chorioamnionitis has both neonatal and maternal benefits. Less known is the ideal postpartum antibiotic regimen - or if postpartum antibiotics are even required at all - needed to decrease febrile morbidity. Current practice has seen a wide range of practice styles ranging from no treatment to antibiotic prophylaxis for up to 48 hours after delivery.

If antibiotics are prescribed, there is good evidence to support one additional dose of antibiotics as compared to 24 hour dosing to decrease the rate of endometritis. Less clear is whether antibiotics are required at all for the properly treated patient with chorioamnionitis who requires a cesarean delivery. One study comparing continued antibiotics versus no-treatment failed to show a difference in the rate of postpartum endometritis. The conclusion from this study was that continuation of preoperative clindamycin and gentamicin in the postoperative period did not reduce the risk of endometritis compared to a single preoperative dose however this study was terminated early due to failure to recruit their stated sample size.

Puerperal endometritis rates vary by mode of delivery but it is known that the rate is lower in vaginal deliveries as compared to cesarean delivery. The patient with chorioamnionitis that requires a cesarean delivery makes an excellent study target. Given the lack of studied protocols, there currently are many acceptable methods for treating the patient with chorioamnionitis. Our proposed study plans to evaluate the two most common methods of treatment to determine the most effective regimen. If post-delivery antibiotics do not show a benefit to these highest risk subjects, it is likely inferred that patients that undergo a vaginal delivery will not require antibiotics as well.

Specific Aims There is conflicting data regarding the necessity of post-delivery antibiotics for patients with chorioamnionitis who undergo cesarean delivery. The primary objective of this study is to determine if postpartum antibiotics are necessary for antepartum treated cases of chorioamnionitis in patients undergoing a cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chorioamnionitis
* Undergoing cesarean section for delivery

Exclusion Criteria:

* Multiple gestations,
* Allergy to beta-lactam antibiotics
* Patients with estimated creatinine clearance (ClCr) less than 70 mL/min
* Maternal fever explained by etiology other than chorioamnionitis
* Inability to comply with the study protocol.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L Shanks, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University, St Louis, Missouri

REFERENCES:
- [Background] Gibbs RS, Dinsmoor MJ, Newton ER, Ramamurthy RS. A randomized trial of intrapartum versus immediate postpartum treatment of women with intra-amniotic infection. Obstet Gynecol. 1988 Dec;72(6):823-8. doi: 10.1097/00006250-198812000-00001. PMID 3186087
- [Background] Sperling RS, Ramamurthy RS, Gibbs RS. A comparison of intrapartum versus immediate postpartum treatment of intra-amniotic infection. Obstet Gynecol. 1987 Dec;70(6):861-5. PMID 3684121
- [Background] Gilstrap LC 3rd, Leveno KJ, Cox SM, Burris JS, Mashburn M, Rosenfeld CR. Intrapartum treatment of acute chorioamnionitis: impact on neonatal sepsis. Am J Obstet Gynecol. 1988 Sep;159(3):579-83. doi: 10.1016/s0002-9378(88)80012-7. PMID 3421256
- [Background] Edwards RK, Duff P. Single additional dose postpartum therapy for women with chorioamnionitis. Obstet Gynecol. 2003 Nov;102(5 Pt 1):957-61. doi: 10.1016/s0029-7844(03)00863-9. PMID 14672470
- [Background] Chapman SJ, Owen J. Randomized trial of single-dose versus multiple-dose cefotetan for the postpartum treatment of intrapartum chorioamnionitis. Am J Obstet Gynecol. 1997 Oct;177(4):831-4. doi: 10.1016/s0002-9378(97)70277-1. PMID 9369828
- [Background] Turnquest MA, How HY, Cook CR, O'Rourke TP, Cureton AC, Spinnato JA, Brown HL. Chorioamnionitis: is continuation of antibiotic therapy necessary after cesarean section? Am J Obstet Gynecol. 1998 Nov;179(5):1261-6. doi: 10.1016/s0002-9378(98)70143-7. PMID 9822512
- [Background] Duff P. Pathophysiology and management of postcesarean endomyometritis. Obstet Gynecol. 1986 Feb;67(2):269-76. doi: 10.1097/00006250-198602000-00021. PMID 3511414

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics
Started | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (6) | 25.3 (6.6) | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 26 | 49
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Paricipants With Endometritis
Description: Endometritis is defined as uterine infection and is diagnosed by maternal temp > 38.0C on two occasions over a 4 hour period or any temp > 39.0C after delivery > 12 hours after delivery. Endometritis will be managed per currently accepted endometritis protocol - (Amp 2 gQ6, Gentamicin 5 mg/kg q24, Clindamycin 900 mg q8).
Time Frame: 7 days post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics
Number analyzed (Participants) | 41 | 39
Participants | 4 | 3

2. Secondary Outcome: Number of Participants With Infection-related Complications
Description: Infection related complications will include common complications attributed to infections there are not the primary outcome (endometritis). This will include infections of the wound and pelvic abscesses.
Time Frame: 7 days post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics
Number analyzed (Participants) | 41 | 39
Participants | 7 | 2

3. Secondary Outcome: Duration of Hospital Stay After Cesarean Delivery
Description: This is the duration of hospital stay (in days) after their cesarean delivery.
Time Frame: Up to 7 Days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics
Number analyzed (Participants) | 41 | 39
days | 4 [4 to 4] | 4 [3 to 4]

ADVERSE EVENTS:
Arm/Group | Postpartum Antibiotics | No Postpartum Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes